CLINICAL TRIAL: NCT06030063
Title: The Society for Obstetric Anesthesia and Perinatology Research Network General Anesthesia Registry
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 2000033638
Record Dates: First submitted 2023-08-16; First posted 2023-09-08 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Cesarean Delivery; General Anesthesia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The SOAP registry is a prospective, multicenter, electronic registry. The goal is to investigate the indications, mode of airway management, predisposing factors, and obstetric and anesthetic outcomes of pregnant patients who receive general anesthesia for cesarean delivery.

DETAILED DESCRIPTION:
This is a central repository with data from 25-40 participating SOAP institutions/hospitals.

The primary and secondary aims of this study are as follows:

1. To determine the institutional factors associated with rates of general anesthesia for cesarean delivery
2. To perform a descriptive analysis of characteristics of general anesthesia for cesarean delivery cases
3. To determine maternal and anesthetic predictors of difficult intubation

Data will be collected from each participating SOAP institution. Institutional data will include information on the characteristics of the institution such as maternal level of care, numbers of lives birth, staffing models, etc. This data will be collected prior to subjects being enrolled into the registry and again at the registry closure to look at intuitional changes over time.

Inclusion into the registry is based on the following criteria:

1. Pregnant women who have had a general anesthetic for Cesarean delivery
2. 15-55 years old

The general anesthesia registry will collect data on subject demographics in a deidentified manner, including characteristics of the birth and delivery, gestational age, maternal morbidities, and anesthetic management.

The granular detail requested in the registry database will help to better understand the nuances of how and why decisions are made about proceeding with general anesthesia in these cases, and once done, how to implement this clinical course. As not all of these data points are routinely recorded in the medical record, optimal data capture requires the treating anesthesiologist to complete the registry entry as soon as possible after conclusion of patient care.

Data will be collected for approximately 5 years and maintained indefinitely. Data is entered into a Yale REDCap registry and will not contain subject identifiers. An estimated 5000 subjects will be enrolled into the data repository. This is based on a published report of 45 institutions' data investigating a subtopic of this question (15 years yielding 15,000 general anesthetics).

ELIGIBILITY:
Inclusion Criteria:

-Pregnant women aged 15-55 who have had a general anesthetic for Cesarean delivery

Ages: 15 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: The subject population will reflect the diverse populations of the participating hospitals. The subject population will include pregnant women aged 15-55 years old who have a general anesthetic during their cesarean delivery. Non-English-speaking subjects will be included.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Rates of General Anesthesia for Cesarean Delivery | Up to 5 years
  The rates of general anesthesia for cesarean delivery among the institutions in the cohort will be assessed. Descriptive analyses of etiologies of and management of general anesthetics for cesarean delivery will also be performed.
Univariate Association Between Facility Type and the Rate of General Anesthesia for Cesarean Delivery | Up to 5 years
  The association between facility type- non-academic affiliated private vs. academic affiliated private vs. military vs. academic (reference)- with a difference in rates of general anesthesia for cesarean delivery will be assessed.
Univariate Association Between SOAP Center of Excellence Designation and the Rate of General Anesthesia for Cesarean Delivery | Up to 5 years
  The association between SOAP center of excellence designation- yes (reference) vs. no- with a difference in rates of general anesthesia for cesarean delivery will be assessed.
Univariate Association Between Maternal Level of Care and the Rate of General Anesthesia for Cesarean Association | Up to 5 years
  The association between maternal level of care- I vs. II vs. III vs. IV (reference)- with a difference in rates of general anesthesia for cesarean delivery will be assessed.
Univariate Association Between Annual Live Births and the Rate of General Anesthesia for Cesarean Delivery | Up to 5 years
  The association between increased numbers of annual live births (continuous variable) and a difference in rates of general anesthesia for cesarean delivery will be assessed.
Univariate Association Between Obstetric Anesthesiologist Coverage and the Rate of General Anesthesia for Cesarean Delivery | Up to 5 years
  The association between increased rates of labor and delivery floor coverage by obstetric anesthesiologists (continuous variable) and a difference in rates of general anesthesia for cesarean delivery will be assessed.
Univariate Association Between Institutional Policies for Labor Epidural Management and the Rate of General Anesthesia for Cesarean Delivery | Up to 5 years
  The association between the presence of institutional policies for labor epidural management- yes (reference) vs. no- and a difference in rates of general anesthesia for cesarean delivery will be assessed.

SECONDARY OUTCOMES:
Rates of Difficult Intubation Among Women Undergoing General Anesthesia for Cesarean Delivery | Up to 5 years
  Among the cohort of general anesthetics for cesarean delivery, the incidence of difficult intubation will be determined.
Univariate Association Between Mallampati Score and the Risk of Difficult Intubation | Up to 5 years
  The association between increased Mallampati score- I or II (reference) vs. III vs. IV- and a difference in risk of difficult intubation will be assessed.
Univariate Association Between Neck Mobility and the Risk of Difficult Intubation | Up to 5 years
  The association between neck mobility- full (reference) vs. limited vs. poor and a difference in risk of difficult intubation will be assessed.
Univariate Association Between Neck Circumference and the Risk of Difficult Intubation | Up to 5 years
  The association between neck circumference- thin or average (reference) vs. thick and a difference in risk of difficult intubation will be assessed.
Univariate Association Between Neck Length and the Risk of Difficult Intubation | Up to 5 years
  The association between neck length- long or average (reference) vs. short and a difference in risk of difficult intubation will be assessed.
Univariate Association Between Thyromental Distance and the Risk of Difficult Intubation | Up to 5 years
  The association between thyromental distance- >6.5cm (reference) vs. 3.5-6.5cm vs. <3.5cm and a difference in risk of difficult intubation will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Leffert, MD, Principal Investigator — Yale Univesrity
Locations (35):
- United States (34):
  - University of Arkansas, Little Rock, Arkansas
  - University of California San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - University of Colorado Hospital, Arvada, Colorado
  - Yale University, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - St Lukes Anesthesia Associates of Boise, Boise, Idaho
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Health System, Kansas City, Kansas
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Mercy Hospital St. Louis, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - University of New Mexico, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Northwell Health, Manhasset, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Renaissance School of Medicine Stony Brook University, Stony Brook, New York
  - Duke University Medical Center, Durham, North Carolina
  - Atrium Health Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University o Cincinnati, Cincinnati, Ohio
  - Ohio State University/Wexner Medical Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas-Houston, Houston, Texas
  - Baylor Scott & White Medical Center, Temple, Texas
  - University of Virginia, Charlottesville, Virginia
- Royal Columbian Hospital & University of British Columbia, New Westminster, Canada